CLINICAL TRIAL: NCT02194972
Title: Study of Soluble Dietary Fiber on Colonic Transit Time and Clinical Symptoms in Adults With Slow-transit Constipation
Brief Title: Clinical Effects of Soluble Dietary Fiber Supplementation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Nanjing PLA General Hospital, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011NLY42
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2014-07

CONDITIONS: Hypomotility; Constipation
Keywords: constipation; colon transit time; gut microbiota; soluble dietary fiber; disturbance of gut microbiota in constipation
MeSH Terms: conditions — Constipation | interventions — Pectins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- soluble dietary fiber (Experimental): pectin, a kind of soluble dietary fiber
  Interventions: Drug: Pectin
- Placebo (No Intervention): Placebo

INTERVENTIONS:
Drug: Pectin — pectin （Andeli Ltd. Yantai, China）, 24g/d for 4weeks
  Other Names: soluble dietary fiber
  Arms: soluble dietary fiber

SUMMARY:
The purpose of this study is to investigate the effect of pectin, a kind of soluble dietary fiber, on colonic transit time, clinical symptoms and the gut microbiota in adults with slow-transit constipation.

DETAILED DESCRIPTION:
Patients were randomized to receive either pectin or placebo. Treatment consisted of 4 weeks supplementation with pectin (fiber group) or placebo. We evaluated the colonic transit time, constipation symptoms and fecal bacterial population in two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients(age≧18y)
* Admitted for slow-transit constipation were considered eligible

Exclusion Criteria:

* Mental disorders
* Cancer
* Inflammatory bowel disease

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
efficacy: intestinal transit time | four weeks after inclusion
  colonic transit time

SECONDARY OUTCOMES:
efficacy: clinical symptoms | four weeks after inclusion
  Wexner constipation score
efficacy: gut microbiota | four weeks after inclusion
  real-time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Tao Gao, M.D., Principal Investigator — Nanjing PLA General Hospital